CLINICAL TRIAL: NCT02833519
Title: Effect of Group Exercise on Mental Wellbeing Among Pregnant Women at Risk of Perinatal Depression: A Randomized Controlled Clinical Trial
Brief Title: Exercise and Wellbeing: The Effect of Group Exercise on Mental Wellbeing Among Pregnant Women
Acronym: EWE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Hanne Kristine Hegaard, Midwife, PhD, Associate professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Rigshospitalet, Denmark
Record Dates: First submitted 2016-05-19; First posted 2016-07-14 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Depression
Keywords: pregnant women; exercise; depression; anxiety
MeSH Terms: conditions — Depression; Motor Activity; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control group (No Intervention): Standard care, mentally vulnerable women
- group exercise (Active Comparator): Supervised Group training
  Interventions: Behavioral: group exercise

INTERVENTIONS:
Behavioral: group exercise — 1. Group training supervised by Physiotherapists from Copenhagen University Hospital, Rigshospitalet. 70 minutes sessions twice a week for 12 weeks.
     The training consists of 10 minutes of warm up (Borg scale 7-10), 20 minutes of fitness training on exercise bike, tread mill or cross-trainer (Borg scale 11-15), 25 minutes of muscle training and 15 minutes stretching/relaxation, (Borg scale 6).
     The intensity of the training follows national recommendations on physical activity for pregnant women, which recommends moderate physical activity or more depending on the pregnant woman's fitness level prior to pregnancy.
  2. The pregnant women´s general practitioners are informed about the intervention and who is participating in the project.
  3. A weekly supportive email.
  Arms: group exercise

SUMMARY:
The purpose of this study is to examine the effect of supervised group exercise on mental wellbeing and signs of depression among pregnant women at risk of perinatal depression in a randomized controlled clinical trial.

The investigators hypothesis is that 70 minutes of supervised group exercise twice a week for 12 weeks by pregnant women at risk of perinatal depression, will improve the participants mental wellbeing and reduce their symptoms of depression.

DETAILED DESCRIPTION:
Pregnant women with a current or a previous history of depression and/or anxiety have a significantly increased risk of perinatal depression and disruptions in the mother-infant attachment. In addition, pregnant women with anxiety and/or depression are at higher risk of preterm birth, low birth weight, and complications during birth.

It is well described that physical exercise in general is associated with psychological well-being and a reduced risk of morbidity and mortality in non-pregnant women. Several studies have documented that physical exercise during pregnancy is associated with health benefits for both infants and mothers. Physical exercise during pregnancy is associated with a lower risk of pregnancy- and delivery related complications such as preeclampsia, gestational diabetes mellitus, low back pain, preterm delivery, emergency caesarean section and postpartum depression, as well as contributing to improved mood.

Nevertheless, in the existing literature there are few and only small studies which have examined the effect of exercise on depression among mentally vulnerable pregnant women.

The aim of this study is to examine the effect of supervised group training for pregnant women with a current or a previous history of depression and/or anxiety.

Patient enrollment. The participants will be recruited from the Department of Obstetrics, Rigshospitalet, Denmark, from July 2016 to March 2019. Participants will be selected on the basis of 1) the information provided by the participants general practitioner and 2) an electronic questionnaire received by email and completed by all pregnant women registered to give birth at Rigshospitalet. The information from the questionnaire is routinely transferred to the pregnant women´s medical records.

The first contact to the participant will be made by phone at about 12-14 weeks of gestation, when, as a part of routine care, all mentally vulnerable pregnant women are contacted by a midwife from the Department of Obstetrics, Rigshospitalet. In this interview, the pregnant woman will be given brief information about the trial. If the woman is interested in further information, written participant information about the trial will be send. If the pregnant woman would like to participate in the project, an appointment for a personal meeting is made, where the participant is given more information about the project before written, informed consent is obtained and randomization can take place.

Data collection and management. Questionnaire number one, baseline data: all participants complete a baseline-questionnaire electronically and data are stored in a secured database.

Questionnaire number two (29-34 weeks of gestation) and questionnaire number three (two months after giving birth): the two questionnaires will be sent to the participants by email and the electronically answered questionnaires are stored in a secured database.

Other data will be obtained from patient records.

Sample size. The calculations have been made based on the primary endpoint, World Health Organisation Five Well-being Index (WHO-5) at 29-34 weeks of gestation. The WHO-5 wellbeing index score ranges from 0-100, where 100 is the best possible wellbeing. The average value measured by the WHO-5 wellbeing index at 10-12 weeks of gestation is 62 points with a standard deviation (SD) of 16. This has previously been assessed among pregnant women at the University Hospital, Rigshospitalet. For the calculations at 29-34 weeks of gestation we will use the SD observed at 10-12 weeks of gestation. The investigators expect that the effect of the intervention causes a 10 point higher WHO-5 index score in the intervention group than in the control group at gestational week 29-34, which is clinically significant ("Guide to the well-being index: WHO-5", Danish Health Authority).

It is estimated that 50% of the participants will be following the program for at least 75% of the sessions (high participation, 19-24 sessions) while 35% will be following 50-75% of the sessions (moderate participation, 12-18 sessions) and 15% will be following less than half of the sessions (low participation). The investigators expect that high participation in the training course will lead to an increase of 10 points in the WHO-5 wellbeing index, that moderate participation in the training course will lead to an increase of 7 points, while low participation will lead to an increase of 2 points, all compared to the control group.

This will lead to an average value in the intervention group which is 7.75 points (0.50 x 10 + 0.35 x 7 + 0.15 x 2) higher than the average value in the control group.

With a power of 90% and a two-sided significance level of 5%, a difference in wellbeing-level of 7.75 points (SD = 16) in the two groups at 29 - 34 weeks of gestation can be detected by a two-sample t-test with 91 patients in each group.

The investigators expect that it will be necessary to include a total of 300 pregnant women, as the investigators anticipate that 12.5% in each group will drop out because of discomfort or complications related to pregnancy and that 30% of the remaining 130 participants in each group will not answer the questionnaire at 29-34 weeks of gestation, which leaves 91 participants in each group.

Data analysis. The primary data analysis will be performed on the basis of the intention-to-treat principle. The investigators compare baseline data for the two groups with Student's t-test, chi-square test or non-parametric tests. A large proportion of missing values for the outcome variable is expected due to drop out and non-response to the questionnaire. Data will be assumed Missing At Random (MAR) and therefore observed patient characteristics will be used to impute missing data, by means of multiple imputation.

While it is expected that there will be a drop-out of 12.5% in each group, and that some pregnant women only participate in the group training a few times, the investigators will perform a per-protocol analysis of the pregnant women who performed ≥ 75% of all training sessions, in addition to the intention-to-treat analyses.

A pilot study with 9 women in the intervention group and 11 women in the control group, will be carried out from April - June 2016.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with depression and/or anxiety requiring treatment within the last ten years, and/or intake of antidepressants in the last three months before conception and/or during pregnancy.
* Age ≥18 years
* Singelton pregnancy
* 17th - 22th week of gestation by intervention start
* Appropriate Danish language skills
* Written informed consent

Exclusion Criteria:

* Age <18 years
* Multiple pregnancies
* Abuse problems
* Eating disorders
* Women who have been diagnosed with malformations or chromosomal disorder in the fetus
* Pelvic instability problems in earlier pregnancy (diagnosed by physiotherapist or doctor)
* Severe obstetric complications.

Withdrawal criteria. Participants will be withdrawal from the study after randomization, if one or more of the following criteria are met:

* Occurred pelvic instability
* Preeclampsia
* Vaginal bleeding
* Other factors indicating an increased risk of preterm birth.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-08; Primary Completion 2019-09-09 (Actual); Study Completion 2019-09-09 (Actual)

PRIMARY OUTCOMES:
World Health Organisation Five Well-being Index (WHO-5). | 29th-34th week of gestation
  Psychological well-being will be measured by the World Health Organisation Five Well-being Index (WHO-5) (mean and SD) or (median and range). Please see the published study protocol Broberg et al. Trials (2017) 18:210.

SECONDARY OUTCOMES:
Edinburgh Postnatal Depression Scale (EPDS) | 29th-34th week of gestation and 2 months after delivery
  Symptoms of depression measured by Edinburgh Postnatal Depression Scale (EPDS) will be defined as a cutoff score ≥13 and a cutoff score ≥10. Please see the published study protocol Broberg et al. Trials (2017) 18:210.
The 12-item General Health Questionnaire (GHQ-12) | 29th-34th week of gestation and 2 months after delivery
  Functional ability will be measured by the 12-item General Health Questionnaire (GHQ-12) (mean and SD) or (median and range). Please see the published study protocol Broberg et al. Trials (2017) 18:210.
Spielbergers State Anxiety Inventory (STAI) | 29th-34th week of gestation and 2 months after delivery
  Clinical symptoms of anxiety will be measured by Spielbergers State Anxiety Inventory (STAI) (mean and SD) or (median and range). Please see the published study protocol Broberg et al. Trials (2017) 18:210.
Pittsburgh Sleep Quality Index (PSQI) | 29th-34th week of gestation and 2 months after delivery
  Sleep quality and sleep disturbances will be measured by the Pittsburgh Sleep Quality Index (PSQI) (mean and SD) or (median and range). Please see the published study protocol Broberg et al. Trials (2017) 18:210.
Percentage of participants with sick leave | 29th-34th week of gestation
  Percentage of participants with sick leave, no matter cause. Please see the published study protocol Broberg et al. Trials (2017) 18:210.
Antenatal contacts | 2 weeks post partum
  Antenatal contacts measured as number of scheduled and unscheduled visits with obstetric doctors and midwifes
Hospitalization, length of stay | 2 weeks post partum
  The duration of hospitalization will be measured in days (mean and SD). Please see the published study protocol Broberg et al. Trials (2017) 18:210.
Percentage of participants with respectively spontaneous onset of labor or inducted labor | 2 weeks post partum
  Will be measured as spontaneous onset of labor or induced labor. Please see the published study protocol Broberg et al. Trials (2017) 18:210.
Use of epidural anaesthesia | 2 weeks post partum
  Use of epidural anaesthesia during delivery, yes or no. Please see the published study protocol Broberg et al. Trials (2017) 18:210.
Duration of labor | 2 weeks post partum
  Duration of labor will be measured in hours. Please see the published study protocol Broberg et al. Trials (2017) 18:210.
Mode of delivery. Percentage of participants with respectively spontaneous delivery, vacuum extraction or cesarean section | 2 weeks post partum
  Respectively spontaneous delivery, vacuum extraction or cesarean section. Please see the published study protocol Broberg et al. Trials (2017) 18:210.
Birth weight in kilograms | 2 weeks post partum
  Birth weight in kilograms, mean and SD. Please see the published study protocol Broberg et al. Trials (2017) 18:210.
Birth length in centimeters | 2 weeks post partum
  Birth length in centimeters, mean and SD. Please see the published study protocol Broberg et al. Trials (2017) 18:210.
World Health Organisation Five Well-being Index (WHO-5). | 2 months after delivery
  Five Well-being Index (WHO-5) (mean and SD) or (median and range). Please see the published study protocol Broberg et al. Trials (2017) 18:210.
Consultations by telephone | 2 weeks post partum
  Measured as number of telephone consultations

CONTACTS AND LOCATIONS:
Overall Officials: Hanne K Hegaard, PhD, Principal Investigator — Department of Obstetrics, The Juliane Marie Centre for Women, Children and Reproduction, Copenhagen University Hospital, Rigshospitalet
Locations (1):
- Hanne Kristine Hegaard, Department of Obstetrics, The Juliane Marie Centre for Women, Children and Reproduction, Copenhagen University Hospital, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Broberg L, Tabor A, Rosthoj S, Backhausen M, Frokjaer VG, Damm P, Hegaard HK. Effect of supervised group exercise on psychological well-being among pregnant women with or at high risk of depression (the EWE Study): A randomized controlled trial. Acta Obstet Gynecol Scand. 2021 Jan;100(1):129-138. doi: 10.1111/aogs.13982. Epub 2020 Sep 15. PMID 32862425
- [Derived] Broberg L, Backhausen M, Damm P, Bech P, Tabor A, Hegaard HK. Effect of supervised exercise in groups on psychological well-being among pregnant women at risk of depression (the EWE Study): study protocol for a randomized controlled trial. Trials. 2017 May 5;18(1):210. doi: 10.1186/s13063-017-1938-z. PMID 28476136